CLINICAL TRIAL: NCT00696553
Title: Randomized Trial of Specialized Nutrition Therapy (SNT) Versus SNT Plus Resistance Training (RT) in Head and Neck Cancer Patients Undergoing Concurrent Chemo-Radiation Therapy (CCR)
Brief Title: Nutrition and Resistance Training in Head and Neck Cancer
Acronym: ELAF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Lance Armstrong Foundation (Other); Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Heidi J. Silver, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 080219
Record Dates: First submitted 2008-06-02; First posted 2008-06-12 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Nutritional Status; Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- B1 (Active Comparator): Nutrition
  Interventions: Other: Tailored Nutrition Intervention
- B2 (Experimental): Nutrition plus Exercise
  Interventions: Behavioral: Nutrition plus Exercise

INTERVENTIONS:
Other: Tailored Nutrition Intervention — Provision of individualized nutrition counseling and nutrition support using oral liquid nutrition supplements and/or liquid enteral supplements
  Arms: B1
Behavioral: Nutrition plus Exercise — Nutrition plus Exercise
  Arms: B2

SUMMARY:
To test the effects of nutrition versus nutrition with resistance exercise on muscle mass loss, fatigue and outcomes of concurrent chemo radiation.

ELIGIBILITY:
Inclusion Criteria:

* Stage 3 or 4 HNC

Exclusion Criteria:

* Previous Cancer

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
muscle mass loss | 6 months

SECONDARY OUTCOMES:
fatigue | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Heidi J Silver, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States